CLINICAL TRIAL: NCT04562701
Title: Relationship Between Hamstring Length and Gluteus Maximums Strength With and Without Normalization in Mechanical Low Back Pain
Brief Title: Relationship Between Hamstring Length and Gluteus Maximums in Mechanical Low Back Pain
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: Prof.Dr Nadia Abdelazim fayaz (Unknown); Walaa Mohsen Mohamed (Unknown); Nagy Sabet (Unknown); Hamada Ahmad Hamada (Unknown)
Responsible Party: Principal Investigator, Nasr Awad Abdelkader Othman, Lecturer, Cairo University
Other Study IDs: P.T.REC/012/002047
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Mechanical Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to determine the correlation between hamstring length and gluteus maximus strength with and without normalization in patients with mechanical low back pain

DETAILED DESCRIPTION:
seventy-three patients diagnosed as mechanical low back pain. Firstly, gluteus maximus (GM) strength was measured isometrically as a force (kg) and then converted to torque (Nm). GM strength was normalized for body weight and height using the following formula: % (body weight × h) = torque (N × m) ×100 / body weight (N) × h (m), then assessment of hamstring length flexibility using the active knee extension method.

Data was collected and the correlation was determined.

ELIGIBILITY:
Inclusion criteria:

* Patients diagnosed as mechanical low back pain (MLBP) with very high grade mechanical inflammatory low back pain (MIL) index.
* Age ranged from 18 to 40 years.
* Body mass index ranged from 25 to 30 kg/m2

Exclusion Criteria:

* History of previous fractures, surgeries, malignancies, trauma, rheumatoid arthritis, spondylosis, and spondylolisthesis.
* History of lower limb injuries in the last six months before the study.
* Inability to correctly produce maximal Gluteus Maximus contraction in a pain-free ROM.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: * Male and female patients
  * Age ranged from 18-40 years
  * Body mass index ranged from 25-30 kg/m2
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2020-01-05 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Gluteus muscle torque | 20 minutes
  The gluteus maximus strength was evaluated by using hand-held dynamometer (HHD). The patient was asked to lie in the prone position. Belt was used to support the pelvis, then the patient was asked to maximally extend the hip joint with the knee joints flexed to 90°). Resistance belt (non-elastic strap) was placed 15 cm above the knee joint above popliteal fossa with the Hand-held dynamometer below it. Each subject was instructed to perform maximal isometric hip extension for 5 seconds. Measurement was done three times, with 2-minutes rest between trials. Subject's hand was places behind waist to control the substitute motions of arm or hand. The peak force for each trial was recorded, and the average value was calculated
Hamstring length | 20 minutes
  Patient was positioned supine with the non-tested limb flat with knee extended and supported with strap over the mid-thigh to eliminate any substitutive movement. An another strap was rapped over the pelvis for fixation, to maintain 90 degrees of the hip joint, a wooden frame was then placed on the plinth in line with the participant's anterior superior iliac spine of the pelvis. The participant was asked to flex the hip of the test leg so that their thigh touching the wooden apparatus all over test time

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Giza, Egypt